CLINICAL TRIAL: NCT07175870
Title: Comparison of Clinical Outcomes Between Preoperative and Postoperative Revascularization in Coronary Heart Disease Patients With Time-Sensitive NOn-Cardiac Surgery: A Multicenter Pragmatic Randomized Controlled Trial (CHRONOS-PCI)
Brief Title: Preoperative vs Postoperative Revascularization in Coronary Heart Disease Patients Undergoing Time-Sensitive Non-Cardiac Surgery (CHRONOS-PCI)
Acronym: CHRONOS-PCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-304
Record Dates: First submitted 2025-09-07; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease; Noncardiac Surgery
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery-First Strategy (Postoperative Revascularization) (Experimental): Patients with coronary heart disease scheduled for time-sensitive non-cardiac surgery. The surgery will be performed in a hybrid operating room. If an acute coronary event occurs intraoperatively, standby PCI will be performed immediately. Elective PCI may also be performed postoperatively if clinically indicated.
  Interventions: Procedure: Preoperative PCI followed by delayed non-cardiac surgery ~3 months later
- PCI-First Strategy (Preoperative PCI with Delayed Surgery) (Active Comparator): Patients with coronary heart disease scheduled for time-sensitive non-cardiac surgery. Participants will undergo PCI first, followed by non-cardiac surgery approximately 3 months later, according to current guideline recommendations for elective surgery after PCI.
  Interventions: Procedure: Non-cardiac surgery followed by postoperative PCI

INTERVENTIONS:
Procedure: Non-cardiac surgery followed by postoperative PCI — Patients undergo the planned time-sensitive non-cardiac surgery first in a hybrid operating room, with PCI standby available in case of an intraoperative acute coronary event. If such an event occurs, immediate PCI will be performed. Additional PCI will be performed postoperatively if clinically indicated.
  Arms: PCI-First Strategy (Preoperative PCI with Delayed Surgery)
Procedure: Preoperative PCI followed by delayed non-cardiac surgery ~3 months later — Patients undergo PCI first. The planned non-cardiac surgery will then be performed approximately 3 months after PCI, in accordance with current guideline recommendations for the timing of non-cardiac surgery following PCI.
  Arms: Surgery-First Strategy (Postoperative Revascularization)

SUMMARY:
To compare the safety and efficacy of preoperative versus postoperative revascularization strategies in patients with coronary heart disease undergoing time-sensitive non-cardiac surgery.

DETAILED DESCRIPTION:
1. Study overview This study is a prospective, open-label, randomized, multicenter trial to evaluate the safety and efficacy of preoperative versus postoperative revascularization strategies in patients with coronary heart disease undergoing time-sensitive non-cardiac surgery.

   The primary hypothesis is that the postoperative (surgery-first) revascularization strategy will show a non-inferior rate of major adverse cardiovascular events (MACE) at 180 days after randomization compared with the preoperative (revascularization-first) strategy.
2. Study population and sample size calculation Based on previous data, the 180-day incidence of MACE was approximately 5.5% in patients undergoing postoperative revascularization and 5.7% in those undergoing preoperative revascularization. Using a non-inferiority margin (delta) of 4%, a two-sided type I error rate (α) of 0.05, and a power of 78%, a total of 140 patients (70 in each group) will be enrolled. An attrition rate of 10% was considered.

   * Primary endpoint: MACE at 180 days after randomization, defined as a composite of all-cause death, myocardial infarction, and any repeat revascularization.
   * Design: Non-inferiority, delta = 4%.
   * Sampling ratio: 1:1 (surgery-first vs. revascularization-first).
   * Type I error (α): Two-sided 0.05.
   * Accrual time: 3 years.
   * Total time: 3.5 years (3 years accrual + 6 months follow-up).
   * Assumption: MACE 5.5% vs. 5.7% in surgery-first and revascularization-first groups, respectively.
   * Statistical power (1-β): 78%.
   * Primary statistical method: Farrington-Manning non-inferiority test for binary outcomes.
   * Potential withdrawal rates: 10%.
   * Stratification in randomization: Randomization will be stratified according to (1) the estimated cardiovascular risk of the non-cardiac surgery and (2) the bleeding risk of the surgery.
3. Research materials and treatment strategies

   * Surgery-first group: Patients will undergo the time-sensitive non-cardiac surgery first. Coronary revascularization (PCI) will be performed after surgery.
   * Revascularization-first group: Patients will undergo coronary revascularization (PCI) prior to the non-cardiac surgery, according to guideline-based recommendations and operator judgment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of coronary heart disease with non-emergent indication for PCI confirmed by coronary angiography：

  * Non-ST-elevation acute coronary syndrome (NSTE-ACS) at low or intermediate ischemic risk
  * Chronic coronary syndrome (CCS) with one of the following anatomical characteristics (see Appendix 1 for definition):

    1. Moderate or severe stenosis of the left main coronary artery
    2. Multivessel disease involving the ostium of the left anterior descending artery
    3. Three-vessel disease with ≥70% stenosis in each major epicardial vessel
* Indication for time-sensitive non-cardiac surgery
* Planned non-cardiac surgery under general anesthesia in the following surgical departments: thoracic surgery, gastrointestinal surgery, colorectal surgery, hepatobiliary and pancreatic surgery, or gynecology
* For patients with malignant tumors requiring time-sensitive surgery: written informed consent confirming understanding and acceptance that, if randomized to the "PCI-first" group, their tumor surgery will be delayed until 90±14 days after PCI, with acknowledgement of potential risks (e.g., tumor progression, change in resectability)
* Ability to understand the study requirements and sign written informed consent in the language provided by the research team

Exclusion Criteria:

* Age >80 years
* Severe thrombocytopenia (platelet count <50×10⁹/L)
* Cardiogenic shock, severe heart failure (NYHA class IV, Killip class IV, or LVEF ≤35%), malignant arrhythmias (including cardiac arrest, asystole, ventricular fibrillation, or sustained ventricular tachycardia), or other life-threatening conditions requiring resuscitation
* Moderate-to-severe valvular heart disease, high-grade atrioventricular block, or other severe cardiac/pulmonary dysfunction incompatible with the planned surgery
* Planned surgery with extremely high bleeding risk (e.g., intracranial surgery, spinal surgery, retinal surgery)
* Patients with malignant tumors undergoing non-palliative surgery who are in poor general condition, defined as meeting any of the following:

  1. Karnofsky performance score <60
  2. Eastern Cooperative Oncology Group (ECOG) performance status >2
* Disease stage beyond surgical indications or estimated life expectancy <1 year
* Patients requiring emergency or urgent surgery due to critical illness
* Severe renal dysfunction: serum creatinine >442 μmol/L, GFR ≤30 mL/min/1.73 m², or currently on renal replacement therapy
* Severe hepatic dysfunction: Child-Pugh class C or higher
* Severe uncontrolled systemic infection
* Advanced dementia with significant decline in quality of life requiring full-time care and support
* Systemic thromboembolic disease (e.g., pulmonary embolism) making surgery unsuitable
* Women who are pregnant, breastfeeding, or planning pregnancy during the study period
* Severe, uncontrolled comorbid conditions continuously impairing physiological or psychological function
* Participation in another clinical study within 3 months prior to enrollment
* Any condition judged by the investigator to interfere with participation or study conduct

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | 180 days after the first invasive procedure (non-cardiac surgery or PCI)
  Composite of all-cause death, myocardial infarction, or repeat revascularization

SECONDARY OUTCOMES:
Major Bleeding | 180 days after the first invasive procedure (non-cardiac surgery or PCI)
  Major bleeding defined as Bleeding Academic Research Consortium (BARC) type 2, 3, or 5 bleeding.
All-Cause Mortality | 180 days after the first invasive procedure (non-cardiac surgery or PCI)
  Death from any cause within 180 days after the first invasive procedure (non-cardiac surgery or PCI)
Myocardial Infarction | 180 days after the first invasive procedure (non-cardiac surgery or PCI)
  Incidence of myocardial infarction defined according to the Fourth Universal Definition
Repeat Coronary Revascularization | 180 days after the first invasive procedure (non-cardiac surgery or PCI)
  Need for repeat PCI of target or non-target coronary arteries
Stroke or Transient Ischemic Attack (TIA) | 180 days after the first invasive procedure (non-cardiac surgery or PCI)
  Incidence of ischemic stroke or TIA confirmed by imaging and neurological evaluation.
New-Onset Acute Heart Failure | 180 days after the first invasive procedure (non-cardiac surgery or PCI)
  Acute onset of heart failure symptoms (e.g., dyspnea, edema, fatigue, palpitations) with clinical signs (including but not limited to displaced apical impulse, cardiac murmur, pulmonary rales, peripheral edema, hepatomegaly) and progressive elevation of BNP or NT-proBNP. Patients must require urgent treatment with intravenous diuretics and/or inotropes.
Myocardial Injury After Non-Cardiac Surgery (MINS) | 72 hours after non-cardiac surgery
  For patients with normal preoperative cTnT: elevation of cTnT within 72 hours after surgery, with at least one value above the 99th percentile URL of the assay, showing a rise/fall pattern suggestive of acute injury; For patients with elevated preoperative cTnT: postoperative increase ≥20% or absolute increase ≥14 ng/L above baseline, or ≥5 ng/L increase above previous concentration, with a peak value >20 ng/L, consistent with acute myocardial injury.
Length of Hospital Stay | 180 days after the first invasive procedure (non-cardiac surgery or PCI)
  Total hospital stay during the study period, including intensive care unit stay, calculated from admission to discharge for the index hospitalization and any subsequent readmissions.
Duke Activity Status Index (DASI) | Baseline and 180±30 days after the first invasive procedure
  Comparison of DASI scores at baseline and at 6 months. The score ranges from 0 to 58.2, with higher scores indicating better functional status.
Fried Frailty Index | Baseline and 180±30 days after the first invasive procedure
  Comparison of Fried scores at baseline and at 6 months. Scoring criteria: 1 point is assigned for each criterion met; a total score ≥3 indicates frailty; 1-2 points indicate a pre-frail state; and 0 points indicate a robust (non-frail) health status.
New York Heart Association (NYHA) classification | Baseline and 180±30 days after the first invasive procedure
  The New York Heart Association (NYHA) classification is a widely used system for grading the severity of heart failure symptoms, ranging from Class I (no limitation of physical activity) to Class IV (symptoms present even at rest, with severe limitations). In this study, we compared the distribution of NYHA classes at baseline and at the 6-month follow-up to evaluate changes in patients' functional status over time.
Patient Health Questionnaire-9 (PHQ-9) depression score. | Baseline and 180±30 days after the first invasive procedure
  The total score of the PHQ-9 can be used to assess the severity of depressive symptoms: 0-4 indicates no depression, 5-9 mild, 10-14 moderate, and ≥15 severe. Comparison of PHQ-9 scores at baseline and at 6 months reflects either the progression or improvement of depressive symptoms in patients.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospitalof Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided